CLINICAL TRIAL: NCT03588819
Title: Two Stereotactic MRI-Guided Ablative Adaptive Radiotherapy Treatments for Localized Prostate Cancer (2SMART)
Brief Title: Stereotactic MRI-Guided Radiation for Localized Prostate Cancer
Acronym: 2SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Andrew Loblaw, GU Radiation Oncology Team Lead, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 014-2018
Record Dates: First submitted 2018-07-02; First posted 2018-07-17 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-fraction SABR (Experimental)
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — 26 Gy in 2 fractions to the prostate and DIL dose of up to 32 Gy in 2 fractions of MR-guided SABR delivered 1 week apart

SUMMARY:
This single arm, prospective study will determine the prostate-specific quality of life (QOL) of patients undergoing undergoing a 2 fraction MRI-guided stereotactic ablative body radiation (SABR) protocol. We propose prescribing a prostate dose of 26 Gy in 2 fractions and a dose of up to 32 Gy to the dominant intraprostatic lesion (DIL) in 2 fractions over one week.

DETAILED DESCRIPTION:
Stereotactic Ablative Body Radiation Two weekly fractions of:

13 Gy to whole prostate +/- seminal vesicles AND Up to 16 Gy simultaneous boost to dominant MRI nodule

Treatment Delivery and Quality Assurance Treatment will be delivered on treatment units equipped with with volumetric arc therapy and hexapod couches. Only photons with megavoltage energies of 6 MV will be used. Cone-beam CT imaging will be performed using the implanted fiducials to set up each treatment. Imaging after each fraction of radiation will be performed and the shifts in prostate positioning (as measured by displacement of gold seed fiducials) will be measured and recorded. Also, the total treatment time for each fraction of radiotherapy will be recorded.

Patient Assessments / Follow-up Time zero will be the start of radiotherapy. Baseline and follow-up parameters are as listed in Appendix A. Baseline rectal and urinary function will be recorded. Acute toxicities will be assessed at weeks 1, 4, and 13 and late toxicities will be assessed at month 6 and every 6 months until year 5 using the Common Terminology Criteria Adverse Events, version 4.0. Bloodwork (PSA and testosterone), will be performed at months 3, 6 and every 6 months until year 5. QOL using the Expanded Prostate Cancer Index Composite (EPIC) will be obtained at baseline, weeks 1, 4, 13, month 6 and every 6 months until year 5.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained
2. Men >18 years
3. Histologically confirmed prostate adenocarcinoma (centrally reviewed)
4. Favorable risk prostate cancer, defined as clinical stage T1-2c, Gleason Sum less than or equal to 7, and PSA less than or equal to 20 ng/mL (patients can have only one of T2c, Gleason Sum 7 and PSA 10-20 ng/ml)

Exclusion Criteria:

1. Androgen deprivation therapy (LHRH-agonists or antiandrogens) > 6 mo
2. Prior pelvic radiotherapy
3. Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
4. Diagnosis of bleeding diathesis
5. Large prostate (>90cm3) on imaging
6. Immunosuppressive medications
7. Inflammatory bowel disease
8. Presence of a hip prosthesis
9. Contraindications to having MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2024-01-23 (Estimated); Study Completion 2024-04-23 (Estimated)

PRIMARY OUTCOMES:
QOL | 5 years
  To determine the prostate-specific quality of life (QOL) using the Expanded Prostate Cancer Index Composite (EPIC)

SECONDARY OUTCOMES:
Acute Toxicity | 3months
  Incidence of acute (≤3 months) complications of interest using Common Terminology Criteria for Adverse Events, version 4.0 (CTCAE v4)
Late Toxicity | 5 Years
  Incidence of late (≥6 months) complications of interest (CTCAE v4)
PSA | 5 years
  Proportion of patients with 4 year PSA value < 0.4 ng/ml
Biochemical Recurrance | 5 years
  5 year biochemical failure rates using the Phoenix definition (nadir PSA + 2 ng/mL)
Salvage Therapy | 5 years
  Rate of salvage therapy (ADT, surgery or brachytherapy)
Health Utilities | 5 year
  Health utilities using the EuroQol-5Dimensions (EQ-5D) questionnaire for mobility, usual activities, anxiety/depression, self-care and pain/discomfort.
Health Utilities | 5 year
  Health utilities using the Patient Oriented Prostate Ultility Scale (PORPUS-U) (0=best quality of life to 1=worst quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong WL, Cheung P, Chung H, Chu W, Detsky J, Liu S, Morton G, Szumacher E, Tseng CL, Vesprini D, Davidson M, Ravi A, McGuffin M, Zhang L, Mamedov A, Deabreu A, Kulasingham-Poon M, Loblaw A. To Boost or Not to Boost: Pooled Analyses From 2-Fraction SABR Trials for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2023 Dec 1;117(5):1153-1162. doi: 10.1016/j.ijrobp.2023.06.250. Epub 2023 Jul 5. PMID 37419394